CLINICAL TRIAL: NCT06435819
Title: Advancing Medical Illustration in Patient Education Materials: From Art to Science. Study 2: ECA-enhanced Document Explanation RCT
Brief Title: ECA-enhanced Document Explanation RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Tufts Medical Center (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 427441
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: 3-treatment between-subjects randomized experiment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ECA-2D (Experimental): Participants read a patient education document with the assistance of an embodied conversational agent rendered in 2D on a computer monitor.
  Interventions: Other: Embodied Conversational Agent (ECA)
- ECA-3D (Experimental): Participants read a patient education document with the assistance of an embodied conversational agent in virtual reality.
  Interventions: Other: Embodied Conversational Agent (ECA)
- CONTROL (No Intervention): Participants read a patient education document without assistance.

INTERVENTIONS:
Other: Embodied Conversational Agent (ECA) — A computer-animated character that can explain a medical illustration to laypersons.
  Arms: ECA-2D; ECA-3D

SUMMARY:
The investigators will evaluate a computer-animated character that explains medical illustrations to people, comparing the character to having people understand the illustrations on their own, and also comparing the computer character on a computer display to one in immersive virtual reality. The investigators will determine which method leads to the best understanding and lowest anxiety.

DETAILED DESCRIPTION:
The investigators are developing a new approach to explaining patient education documents and illustrations to patients with varying levels of health literacy, involving the use of Embodied Conversational Agents (ECAs). The investigators will evaluate our ECA-augmented Document Explanation tool to determine whether it improves patient learning relative to traditional static patient education documents. The investigators will conduct a 3-arm randomized between-subjects experiment, in which participants read a patient education document with embedded medical illustration, either unaided (CONTROL), with the assistance of an ECA rendered in 2D on a standard computer monitor (ECA-2D), or with the assistance of an ECA in immersive Virtual Reality (ECA-3D).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Speaks English or Spanish ﬂuently
* Is able to independently consent
* Has adequate corrected vision to read patient education documents

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge | Baseline and 30 minutes
  A multiple-item knowledge test designed to test comprehension of the patient education document
State Anxiety scale from State-Trait Anxiety Inventory | 30 minutes
  Self-report state anxiety scale from the State-Trait Anxiety Inventory. 20 items, 4-point Likert scale. A higher score indicates more severe anxiety with a potential range from 20 to 80.

SECONDARY OUTCOMES:
Satisfaction with illustration | 30 minutes
  Likert items to assess satisfaction with the document and illustration
Reading Effort | 30 minutes
  Likert items to assess perceived effort in reading a document and illustration
Acceptability | 30 minutes
  Likert items to assess acceptability and appropriateness of the illustration

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bickmore, PhD, Principal Investigator — Northeastern University
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Northeastern University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Quantitative measures of comprehension and anxiety will be collected from participants who either have patient education documents explained to them by embodied conversational agents or read the documents themselves. We will create de-identified data sets of all quantitative human subjects data that will be preserved and shared. The purpose for creating this is to allow other investigators access to the data to both validate our findings and to further advance inquiry in the field.
Supporting Information: Study Protocol, ICF
Time Frame: Prior to end of the study.
Access Criteria: Sharing of de-identified human subjects data will be consistent with HIPAA guidelines and the Final NIH Statement on Sharing Research Data. We do not anticipate any limitations on sharing.